CLINICAL TRIAL: NCT05779618
Title: Prevalence of Tongue Anomalies Among Group of Egyptian Children: a Cross-sectional Study
Brief Title: Prevalence of Tongue Anomalies in Egyptian Children
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mostafa Mohamed Elzahaby, Principle investigator, Cairo University
Other Study IDs: 120805
Record Dates: First submitted 2023-03-08; First posted 2023-03-22 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Tongue; Anomaly
Keywords: Tongue anomalies; ankyloglossia; Fissured tongue; Geographic tongue; macroglossia
MeSH Terms: conditions — Congenital Abnormalities; Ankyloglossia; Tongue, Fissured; Glossitis, Benign Migratory; Macroglossia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — observational study, all data collected are binary

SUMMARY:
The purpose of the study is to determine the prevalence of tongue anomalies in a group of Egyptian children and to relate the presence of malocclusion in cases of macroglossia, tongue tie and microglossia.

DETAILED DESCRIPTION:
The tongue is an important and accessible muscle in the oral cavity, it has many functions which includes speech, chewing, swallowing, sucking, control of breathing, growth and developments of the jaws and perception to pain.

Also, many systemic disorders and diseases affect the tongue which makes it a great reflector of the general health.

Tongue anomalies has different frequencies and prevalence between different countries, these differences may be due to geographic, ethnic, gender and age variability, for example a study in Iran in 2003 found that the prevalence of tongue anomalies 34.3%, while another study in Colombia in 2013 found that the prevalence of tongue anomalies on their study population was 79.9%.

The knowledge of the prevalence of tongue anomalies among Egyptian children is missing in the literature which could compromise the quality of dental care, increase the occurrence of orthodontic problems and decrease the chances of early detection of some systemic diseases, since tongue anomalies could help in early determination of some systemic diseases in cases of fissured tongue and geographic tongue as well as early prevention and early intervention of malocclusions and speech defects that might be caused in cases of microglossia, macroglossia and ankyloglossia.

Hence, the knowledge of prevalence of tongue anomalies among Egyptian children can aid in setting a reference which will then help in public health planning and prevention policies.

ELIGIBILITY:
Inclusion Criteria:

* Participants' age between 6-12 years.
* Co-operative child
* Positive participants' acceptance for participation in the study.
* Participants having responsible care giver answered by approval on the previously sent informed consent which describes the aim & importance of the study

Exclusion Criteria:

* Patients with history of significant medical conditions
* Participants undertaken anti-fungal drugs in the previous 12 months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: school children between six to twelve years old
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-03-25 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
prevalence of tongue anomalies | 1 month
  studying the prevalence of tongue anomalies among Egyptian children between 6 to 12 years old

SECONDARY OUTCOMES:
macroglossia, microglossia and ankyloglossia effect on occlusion | 1 month
  detecting the presence or absence of malocclusion in cases of three types of tongue anomalies (ankyloglossia, macroglossia and microglossia)

CONTACTS AND LOCATIONS:
Overall Officials: Randa Abd Al Gawad, Dental PhD, Study Director — Cairo University; Yasmin Yousry, Dental PhD, Study Chair — Cairo University
Locations (2):
- Egypt (2):
  - Aley Ibn Abi Taleb primary school, Cairo
  - Mansheyet Gebril primary school, Cairo

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared via email to other researchers if needed.
Supporting Information: Study Protocol
Time Frame: data will be available starting June 2023 for 1 year

REFERENCES:
- [Background] Rioboo-Crespo Mdel R, Planells-del Pozo P, Rioboo-Garcia R. Epidemiology of the most common oral mucosal diseases in children. Med Oral Patol Oral Cir Bucal. 2005 Nov-Dec;10(5):376-87. English, Spanish. PMID 16264385
- [Background] Suter VG, Bornstein MM. Ankyloglossia: facts and myths in diagnosis and treatment. J Periodontol. 2009 Aug;80(8):1204-19. doi: 10.1902/jop.2009.090086. PMID 19656020
- [Background] Belmehdi A, Harti KE, Wady WE. Ankyloglossia as an oral functional problem and its surgical management. Dent Med Probl. 2018 Apr-Jun;55(2):213-216. doi: 10.17219/dmp/85708. PMID 30152627
- [Background] Avcu N, Kanli A. The prevalence of tongue lesions in 5150 Turkish dental outpatients. Oral Dis. 2003 Jul;9(4):188-95. doi: 10.1034/j.1601-0825.2003.02933.x. PMID 12974518
- [Background] Chang PS, Yen TH, Huang CJ, Yen AM, Chen SL, Tsai AI. Clinical Orodental Anomalies in Taiwanese Children under Age Six: a Study Based on the 1995-1997 National Dental Survey. Biomed Res Int. 2020 Jul 19;2020:2056340. doi: 10.1155/2020/2056340. eCollection 2020. PMID 32766305
- [Background] Rezaei F, Safarzadeh M, Mozafari H, Tavakoli P. Prevalence of Geographic tongue and Related Predisposing Factors in 7-18 Year-Old Students in Kermanshah, Iran 2014. Glob J Health Sci. 2015 Feb 24;7(5):91-5. doi: 10.5539/gjhs.v7n5p91. PMID 26156909